CLINICAL TRIAL: NCT04518059
Title: Assessing Skin Biomarkers for Preclinical Diagnosis of PD and Non-PD Parkinsonism
Brief Title: Misfolded Proteins in the Skin of People With Parkinson's Disease and Other Parkinsonism
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Banner Health (Other); University of Bologna (Other); Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Steven Gunzler, MD, Assistant Professor, Neurology, University Hospitals Cleveland Medical Center
Other Study IDs: 20181189; 1U01NS112010-01 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Parkinsonism; Dementia With Lewy Bodies; Multiple System Atrophy; Progressive Supranuclear Palsy; Corticobasal Degeneration
Keywords: Parkinson disease; Parkinson's disease; dementia with Lewy bodies; multiple system atrophy; progressive supranuclear palsy; corticobasal degeneration; biomarker; parkinsonism; alpha-synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Lewy Body Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Skin and blood samples are collected and used for analysis in the Case Western Reserve University Department of Pathology. Blood samples are obtained for NIH affiliated biobanks BioSEND/PDBP and RUCDR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinsonism Group: Participants with Parkinson's disease (PD), dementia with Lewy bodies (DLB), multiple system atrophy (MSA), progressive supranuclear palsy (PSP), and corticobasal degeneration (CBD)
  Interventions: Procedure: punch skin biopsy
- Control Group: Participants without parkinsonism
  Interventions: Procedure: punch skin biopsy

INTERVENTIONS:
Procedure: punch skin biopsy — An anesthetic medication is injected to numb the areas of skin and two samples of skin are obtained from punch biopsy.

SUMMARY:
The purpose of this study is to determine whether identification of misfolded proteins in the skin will help to determine what sort of parkinsonism someone has. We seek to demonstrate whether someone has a synucleinopathy such as Parkinson's disease (PD), multiple system atrophy (MSA), or dementia with Lewy bodies(DLB), as opposed to a tauopathy such as progressive supranuclear palsy (PSP) or corticobasal degeneration (CBD) or no parkinsonism at all (control).

DETAILED DESCRIPTION:
This is a clinical research study for patients with parkinsonism, including Parkinson's disease, progressive supranuclear palsy, corticobasal degeneration, multiple system atrophy, and dementia with Lewy bodies. Parkinsonism can be difficult to diagnose, especially in the early stages of the disease. Skin punch biopsy could be a useful and way to diagnose and measure the severity of these conditions. Given that there currently is no proven way to determine that someone has a synucleinopathy such as PD and not a tauopathy, this is a novel study that may lead to better ways to diagnose people with parkinsonism. The purpose of the study is to identify changes on a skin punch biopsy, in which small samples of skin are removed and sent to the laboratory for examination. We are seeking to measure the amount of misfolded alpha-synuclein in someone's skin. Participation will last between 1 and 2 years and will involve between 2 and 4 visits. Visits will include a physical examination, questionnaires, a memory test, blood draws and saliva collection, and a single visit for skin punch biopsies. We will also be looking to enroll volunteers to serve as "controls," who do not have any neurological illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years old and age <90 years of age at the time of the baseline visit 1
* Age of diagnosis at least 40 years old for PD, DLB, and PSP and at least 30 years old for MSA
* A confirmed diagnosis of PD, PSP, CBD, MSA, DLB, or healthy control
* Montreal Cognitive Assessment (MoCA) > 10 at the outset of the study

Exclusion Criteria:

* Age 90 or above
* Allergy to local anesthetic
* History of deep brain stimulation (DBS) or other brain surgery prior to Visit 1
* For PD or DLB diagnoses, any other neurodegenerative or central nervous system process that would interfere with examination
* For PD or DLB, history of negative DATscan
* Use of investigational drugs or devices within 60 days prior to baseline visit (except for dietary supplements)
* In control subjects, family history of a neurodegenerative disease in a first degree or second degree blood relative
* History of schizophrenia
* History of antipsychotic medication use or exposure in controls or history of antipsychotic medication leading to parkinsonism (drug induced parkinsonism) in the parkinsonism group
* Blood clotting disorder
* On multiple (more than one) antiplatelet and/or anticoagulant blood thinner medications in combination (except for aspirin if it can be safely held for 1 week)
* Any other medical, psychiatric, or cognitive illness that in the investigator's opinion would interfere with cooperation or ability to undergo the study procedures.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with parkinsonism, Parkinson's disease (PD), dementia with Lewy bodies (DLB), multiple system atrophy (MSA), progressive supranuclear palsy (PSP), and corticobasal degeneration (CBD), and also controls without parkinsonism.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Amount of alpha-synuclein in the skin | Cross-sectional at baseline
  Alpha-synuclein will be measured by RT-QuIC and sPMCA
Change in PSPRS measures of progressive supranuclear palsy (PSP) severity in people with PSP | Baseline, 1 year, and optional 2 year assessment
  Questionnaire and examination. Lower scores are better.
Change in UMSARS measures of multiple system atrophy (MSA) severity in people with MSA | Baseline, 1 year, and optional 2 year assessment
  Questionnaire and examination. Lower scores are better.
Change in Hoehn and Yahr (H&Y) and modified H&Y Scores | Baseline, 1 year, and optional 2 year assessment
  Zero to 5 parkinsonism rating scale score. Lower score is better.
Change in Schwab and England (S&E) Score | Baseline, 1 year, and optional 2 year assessment
  0% to 100% rating scale score. Higher score is better.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Baseline, 1 year, and optional 2 year assessment
  Zero to 30 cognitive rating scale score. Higher score is better.
Change in Epworth Sleepiness Scale (ESS) | Baseline, 1 year, and optional 2 year assessment
  Zero to 24 sleepiness rating scale score. Lower score is better.
Change in Hamilton depression scale | Baseline, 1 year, and optional 2 year assessment
  17 item depression rating scale score. Lower score is better.
Change in Hamilton anxiety scale | Baseline, 1 year, and optional 2 year assessment
  14 item depression rating scale score. Lower score is better.
Change in REM Behavior Disorder Questionnaire | Baseline, 1 year, and optional 2 year assessment
  10 item depression rating scale score. Lower score is better.
Change in blood pressure with orthostatic posture | Baseline, 1 year, and optional 2 year assessment
  Blood pressure from lying down to sitting to standing. Smaller drop in blood pressure is better.
Amount of alpha-synuclein in the blood | Baseline, optional 1 year assessment, and optional 2 year assessment
  Alpha-synuclein will be measured in the blood sample
Change in PDQ-39 | Baseline, optional 1 year assessment, and optional 2 year assessment
  39 item health status questionnaire. Lower is better.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gunzler, MD, Principal Investigator — University Hospitals Cleveland Medical Center and Case Western Reserve University; Chen Shu, PhD, Principal Investigator — University of Alabama at Birmingham; Zerui Wang, MD, PhD, Principal Investigator — Case Western Reserve University; Qingzhong Kong, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals Suburban Health Center, South Euclid, Ohio

IPD SHARING:
Plan to Share IPD: No